CLINICAL TRIAL: NCT01305200
Title: A Randomized Double Blinded Trial of Topical Caphosol to Prevent Oral Mucositis in Children Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Supersaturated Calcium Phosphate Rinse in Preventing Oral Mucositis in Young Patients Undergoing Autologous or Donor Stem Cell Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ACCL1031; NCI-2011-02635 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000695718 (Other: Clinical Trials.gov); ACCL1031 (Other: Children's Oncology Group); COG-ACCL1031 (Other: DCP); ACCL1031 (Other: CTEP); U10CA095861 (NIH)
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2016-11

CONDITIONS: Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; de Novo Myelodysplastic Syndromes; Disseminated Neuroblastoma; Juvenile Myelomonocytic Leukemia; Mucositis; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Previously Treated Childhood Rhabdomyosarcoma; Previously Treated Myelodysplastic Syndromes; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Wilms Tumor and Other Childhood Kidney Tumors; Recurrent/Refractory Childhood Hodgkin Lymphoma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myelomonocytic, Juvenile; Mucositis; Myeloproliferative Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Testicular Neoplasms; Wilms Tumor; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (placebo) (Placebo Comparator): Patients rinse and gargle with placebo over 1 minute QID beginning the first day (about day -7) of the conditioning regimen. Treatment continues until day 20 post-transplantation.
  Interventions: Other: placebo; Other: questionnaire administration; Procedure: quality-of-life assessment
- Arm II (supersaturated calcium phosphate rinse) (Experimental): Patients rinse and gargle with supersaturated calcium phosphate rinse over 1 minute QID beginning on the first day (about day -7) of the conditioning regimen. Treatment continues until day 20 post-transplantation.
  Interventions: Drug: supersaturated calcium phosphate rinse; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: supersaturated calcium phosphate rinse — Mouth rinse
  Other Names: Caphosol
  Arms: Arm II (supersaturated calcium phosphate rinse)
Other: placebo — Mouth rinse
  Other Names: PLCB
  Arms: Arm I (placebo)
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This randomized phase III trial is studying how well Caphosol rinse works in preventing mucositis in young patients undergoing autologous or donor stem cell transplant. Supersaturated calcium phosphate (Caphosol) rinse may be able to prevent mucositis, or mouth sores, in patients undergoing stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if topically administered supersaturated calcium phosphate (Caphosol), rinsed orally four times daily at the initiation of conditioning for hematopoietic stem cell transplantation (HSCT), reduces oral mucositis as demonstrated by a decrease in duration of severe oral mucositis (World Health Organization [WHO] grade 3 or 4), compared to placebo.

SECONDARY OBJECTIVES:

I. To determine whether Caphosol administration, when compared to placebo, reduces oral mucositis as demonstrated by a decrease in incidence of severe oral mucositis (WHO grade 3 or 4); severity of mucositis according to mouth pain categorical rating scale and Oral Mucositis Daily Questionnaire (OMDQ); incidence, total dose, and duration of parenteral opioid analgesic use (morphine equivalents); and incidence and duration of total parenteral nutrition (TPN) administration.

II. To determine whether Caphosol administration, when compared to placebo, reduces the incidence of febrile neutropenia and invasive bacterial infections.

III. To validate a new pediatric measure of oral mucositis termed the Children's International Mucositis Evaluation Scale (ChIMES).

OUTLINE: This is a multicenter study. Patients are stratified according to conditioning regimen (total-body irradiation (TBI) or melphalan vs neither TBI nor melphalan) and hematopoietic stem cell transplantation (HSCT) (autologous vs allogeneic). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients rinse and gargle with supersaturated calcium phosphate rinse over 1 minute four* times daily (QID) beginning on the first day (about day -7) of the conditioning regimen.

ARM II: Patients rinse and gargle with placebo over 1 minute QID* beginning the first day (about day -7) of the conditioning regimen.

NOTE: * Patients who reach WHO grade 3 or 4 mucositis have the option to request a total of 6 rinses daily.

In both arms, treatment continues until day 20 post-transplantation OR until mucositis resolves to WHO grade =< 2 for two consecutive days OR on day 12 in patients who do not experience oral mucositis of at least WHO grade >= 1. Patients are assessed daily by trained healthcare professionals using the Oral Mucositis Daily Questionnaire (OMDQ), the Pain Rating Scale, the WHO Mucositis Scale, and the Children's International Mucositis Evaluation Scale (ChIMES) from day -1 and continuing until day 20. Patients are also observed for the incidence of total dose and duration of parenteral opioid analgesic use, duration of total parenteral nutrition (TPN) administration, febrile neutropenia, and invasive bacterial infections.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing myeloablative autologous or allogeneic hematopoietic stem cell transplantation (HSCT) for any indication
* One or more of the following donor stem cell sources (autologous or allogeneic):

  * Bone marrow
  * Placental blood (umbilical cord blood)
  * Cytokine-mobilized peripheral blood
* Patients eligible for allogeneic HSCT must have one of the following types of donor stem cells:

  * Human leukocyte antigen (HLA)-matched sibling or parent
  * Partially matched family donor (mismatched for a single HLA locus [Class I])
  * Fully matched unrelated marrow or peripheral blood stem cell donor
  * HLA-matched or partially mismatched (at least 4 of 6 match) cord blood (Class I or II)
* Patients expecting to receive any type of myeloablative HSCT conditioning regimen are eligible

  * No non-myeloablative or reduced-intensity conditioning regimens
* Eligible patients must not have received palifermin within 30 days prior to enrollment
* Eligible patients must not have received prior treatment with Caphosol

Exclusion Criteria:

* Females of childbearing potential must have a negative pregnancy test; patients must agree to use an effective birth control method; lactating patients must agree not to nurse a child while on this trial

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 226 (Actual)
Dates: Start 2011-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Treister, MD, Principal Investigator — Children's Oncology Group
Locations (35):
- United States (31):
  - Children's Oncology Group, Arcadia, California
  - City of Hope, Duarte, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Miami Children's Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital-Main Campus, New Orleans, Louisiana
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ny Cancer%, Valhalla, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Royal Childrens Hospital, Herston, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec

REFERENCES:
- [Background] Treister N, Nieder M, Baggott C, Olson E, Chen L, Dang H, Krailo M, August A, Sung L. Caphosol for prevention of oral mucositis in pediatric myeloablative haematopoietic cell transplantation. Br J Cancer. 2017 Jan 3;116(1):21-27. doi: 10.1038/bjc.2016.380. Epub 2016 Nov 22. PMID 27875526
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm III (Enrolled But Not Randomized): Site not randomized
Period: Overall Study
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse) | Arm III (Enrolled But Not Randomized)
Started | 111 | 112 | 3
Completed | 82 | 81 | 0
Not Completed | 29 | 31 | 3
Not completed — Physician Decision | 4 | 6 | 1
Not completed — Withdrawal by Subject | 24 | 21 | 1
Not completed — Ineligible | 1 | 2 | 1
Not completed — Death | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm III (Enrolled Not Randomized): Site not able to randomize.
- Total: Total of all reporting groups
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse) | Arm III (Enrolled Not Randomized) | Total
Number analyzed (Participants) | 111 | 112 | 3 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.75 (5.05) | 13.02 (4.54) | 12.00 (1.73) | 12.88 (4.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 48 | 2 | 104
  Male | 57 | 64 | 1 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 29 | 1 | 55
  Not Hispanic or Latino | 82 | 79 | 2 | 163
  Unknown or Not Reported | 4 | 4 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 4 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 11 | 0 | 23
  White | 87 | 82 | 3 | 172
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 14 | 0 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5 | 4 | 0 | 9
  United States | 105 | 102 | 3 | 210
  Australia | 1 | 5 | 0 | 6
  Puerto Rico | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe Oral Mucositis (WHO Grade 3 or 4)
Description: Mean days of severe (WHO Grade 3 or 4) Mucositis.
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation.
Population: Evaluable patients defined as patients with >= 11 daily WHO assessments.
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 91 | 91
Number of days | 4.5 (4.8) | 4.5 (5)

2. Secondary Outcome: Incidence of Severe Oral Mucositis
Description: Percentage of patients with Severe Oral Mucositis (WHO Grade 3 or 4) per arm.
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation.
Population: Evaluable patients defined as patients with >= 11 daily WHO assessments.
Measure: Number; unit: percent of patients
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 91 | 91
percent of patients | 68 | 63

3. Secondary Outcome: Oral Mucositis Daily Questionnaire (OMDQ)
Description: Area under the curve (AUC) of the Oral Mucositis Daily Questionnaire (OMDQ) subscales
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation
Population: Evaluable patients defined as patients with ≥11 daily WHO assessments.
Measure: Mean (Standard Deviation); unit: units on a scale * day
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 91 | 91
units on a scale * day
  Sleeping | 9.3 (10.9) | 7.3 (9)
  Mouth and Throat Pain | 22.3 (14.8) | 21.4 (14.7)
  Swallowing | 21.4 (15.7) | 19.9 (15.9)
  Drinking | 21.7 (16.3) | 20.6 (17.3)
  Eating | 27.9 (19.4) | 26.6 (20.7)
  Talking | 12.2 (11.5) | 12 (13.2)

4. Secondary Outcome: Incidence of Parenteral Opioid Analgesic Use (Morphine Equivalents).
Description: Opioid Administration = yes
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation.
Population: Total of 210 patients evaluable for this assessment (106 Arm I & 104 Arm II)
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 106 | 104
percentage of participants | 88.7 | 91.3

5. Secondary Outcome: Duration of Parenteral Opioid Analgesic Use (Morphine Equivalents).
Description: Mean days of parenteral opioid analgesic use.
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation.
Population: Total of 210 patients evaluable for this assessment (106 Arm I & 104 Arm II).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 106 | 104
Days | 14.2 (9.5) | 12.5 (8.7)

6. Secondary Outcome: Total Dose of Parenteral Opioid Analgesic Used (Morphine Equivalents).
Description: Morphine equivalent dose in mg/kg/day
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation.
Population: Total of 210 patients evaluable for this assessment (106 Arm I & 104 Arm II).
Measure: Median (Full Range); unit: mg/kg/day of opioid analgesics
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 106 | 104
mg/kg/day of opioid analgesics | 0.4 [0 to 33.2] | 0.3 [0 to 13.4]

7. Secondary Outcome: Incidence of Total Parenteral Nutrition (TPN) Administration.
Description: Total Parenteral Nutrition = yes
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation.
Population: Total of 210 patients evaluable for this assessment (106 Arm I & 104 Arm II).
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 106 | 104
percentage of participants | 78.3 | 72.1

8. Secondary Outcome: Duration of Total Parenteral Nutrition (TPN) Administration.
Description: Mean days of total parenteral nutrition (TPN) administration.
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation.
Population: Total of 210 patients evaluable for this assessment (106 Arm I & 104 Arm II).
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 106 | 104
Number of days | 13.6 (9.9) | 11.4 (8.9)

9. Secondary Outcome: Incidence of Febrile Neutropenia
Description: Fever and Neutropenia = yes
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation.
Population: Total of 210 patients evaluable for this assessment (106 Arm I & 104 Arm II).
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 106 | 104
percentage of participants | 65.1 | 67.3

10. Secondary Outcome: Incidence of Invasive Bacterial Infections
Description: Invasive Bacterial Infection = yes
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation.
Population: Total of 210 patients evaluable for this assessment (106 Arm I & 104 Arm II).
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 106 | 104
percentage of participants | 6.6 | 7.7

11. Secondary Outcome: Severity of Mucositis
Description: Area Under the Curve of Severity of Mucositis. According to mouth pain categorical rating scale ranges 0-10 with higher scores reflecting more severe pain.
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation
Population: Evaluable patients defined as patients with ≥11 daily WHO assessments.
Measure: Mean (Standard Deviation); unit: units on a scale * day
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 91 | 91
units on a scale * day | 45.5 (36) | 44 (35.6)

12. Other Pre Specified Outcome: Ancillary Validation Study of ChIMES
Time Frame: Day -1 (day prior to stem cell infusion) to Day 20 following transplantation.
Population: Analysis is not performed at this time due to no available funding and no human resource allocated to this study.
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Total of 210 patients evaluable for toxicity (106 Arm I & 104 Arm II). Reasons for exclusion from this population include 3 ineligibles, 3 not randomized, 10 off before starting study/treatment.
Arm/Group | Arm I (Placebo) | Arm II (Supersaturated Calcium Phosphate Rinse)
Serious Adverse Events (participants affected / at risk) | 0/106 | 3/104
Other Adverse Events (participants affected / at risk) | 29/106 | 22/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Placebo) (N=106) | Arm II (Supersaturated Calcium Phosphate Rinse) (N=104)
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Placebo) (N=106) | Arm II (Supersaturated Calcium Phosphate Rinse) (N=104)
Allergic reaction (Immune system disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 12 | 8
Neutrophil count decreased (Investigations) | 0 | 1
Oral pain (Gastrointestinal disorders) | 16 | 13
Pain (General disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other